CLINICAL TRIAL: NCT02143427
Title: Treatment of Children With Peer Related Aggressive Behavior With the Computer Based Treatment Program ScouT - a Randomized Controlled Trial
Brief Title: Treatment of Children With Peer Related Aggressive Behavior (ScouT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, Anja Goertz-Dorten, PhD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ScouT-Study 1
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Oppositional Defiant Disorder
Keywords: social skills training,; computer based,; social competence training,; Oppositional Defiant Disorder; peer related aggressive behavior; randomized controlled trial
MeSH Terms: conditions — Oppositional Defiant Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Skills Training (Experimental): Social Skills Training child-focused and subsequent social competence training which combines patient- and parent-/teacher and peer-focused interventions
  Interventions: Behavioral: Social Skills Training
- Treatment Program with techniques to activate resources (Active Comparator): Treatment Program with techniques to activate resources of the child and subsequent Social Skills Training child-focused
  Interventions: Behavioral: Treatment Program with techniques to activate resources

INTERVENTIONS:
Behavioral: Social Skills Training — Behavioral: computer-based Treatment Program for Children with Aggressive Behavior 16 sessions with the child aiming at the reduction of peer related aggressive behavior via social skills training. Additionally up to 2 sessions with relatives of the child in most cases with the parents and subsequent Treatment Program for Children with Aggressive Behavior 16 sessions with the child aiming at the reduction of peer related aggressive behavior via social skills training. Additionally up to 6 sessions with relatives of the child in most cases with the parents.
  Arms: Social Skills Training
  Arms: Social Skills Training
Behavioral: Treatment Program with techniques to activate resources — Behavioral: Treatment Program with techniques to activate resources 16 sessions with the child aiming at the reduction of peer related aggressive behavior via activate resources. Additionally up to 2 sessions with relatives of the child in most cases with the parents and subsequent computer based Treatment Program for Children with Aggressive Behavior 16 sessions with the child aiming at the reduction of peer related aggressive behavior via social skills training.
  Arms: Treatment Program with techniques to activate resources of the child and subsequent Social Skills Training
  Arms: Treatment Program with techniques to activate resources

SUMMARY:
The efficacy of the computer based Treatment Program for Children with Aggressive Behaviour (Soziales computerunterstütztes Training für Kinder mit aggressivem Verhalten, ScouT) which is a child focused social competence training delivered in an individual format will be evaluated in a randomized controlled trial with children aged 6 to 12 years with peer-related aggressive behaviour.

DETAILED DESCRIPTION:
The German computer based Treatment Program for Children with Aggressive Behaviour (Soziales computerunterstütztes Training für Kinder mit aggressivem Verhalten, ScouT) aims at the therapy of children aged 6 to 12 years with peer-related aggressive behaviour, which results in a persistent impairment of the relationships to other children. Contrary to other treatment approaches, this intervention aims at the individual treatment of problem maintaining and moderating factors of aggressive behaviour. Depending on the individual problem maintaining factors the treatment aims to modify social cognitive information processing, social problem solving and behavioral social skills.

Methods: The efficacy will be tested in a randomized control group design with n=140 children. N=70 children will be treated in the first treatment phase (pre- to post1-assessment) of 16 weekly child-focused sessions with the treatment modules of ScouT. In the second treatment phase (post1- to post2- assessment) those children with sustained severe peer related aggressive behavior receive the comprehensive Treatment Program for Children with Aggressive Behaviour (Therapieprogramm für Kinder mit aggressivem Verhalten, THAV) which is a social competence training which combines patient- and parent-/teacher and peer-focused interventions with 16 child sessions and 6 parent-/teacher sessions. Those children with no severe peer related aggressive behavior receive 2 booster sessions of ScouT within a 16 week period.

The control group of n=70 children will receive in the first treatment phase (pre- to post1-assessment) an alternative child-focused intervention with a supportive Treatment Programm including techniques to activate resources of the child (Supportive Therapie zur Aktivierung von Ressourcen bei Kindern, STARK) with 16 weekly sessions. In the second treatment phase (post1- to post2- assessment) those children with sustained severe peer related aggressive behavior receive 16 weekly child-focused sessions with the treatment modules of ScouT . Those children with no severe peer related aggressive behavior receive 2 booster sessions of STARK within a 16 week period.

A follow-up assessment is conducted 12 months after post2-assessment. Outcome parameters are aggressive behaviour und comorbid symptoms as well as problem maintaining factors, psychosocial functioning, family burden, self-esteem and treatment satisfaction as rated by clinicians, parents, or teachers. Additionally problem solving is assessed by a newly developed problem-solving test. Moreover, variables of the treatment process are assessed. Additionally treatment process parameters are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 - 12 years
* IQ>= 80
* Diagnoses (ICD-10): F91, F92, F90.1
* Elevated symptom score in the parent rated Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV) with Stanine ≥ 7 at pre-assessment
* Often conflicts with other children (clinical rating)
* Impaired social relationships / activities
* Parents agree in randomization (clinical rating) in medicated children no planned change of the medication

Exclusion Criteria:

* Other disorder is dominating
* Other active psychotherapy
* Severe mental disorder of the parents

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
total score for peer related aggression in the Questionnaire for Aggressive Behavior of Children (FAVK) parent rating | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The Questionnaire for Aggressive Behavior of Children (FAVK) is a newly developed parent rating scale which assesses several factors of peer related aggression: (1) disturbance of social cognitive information processing, (2) disturbance of social problem solving and social skills, (3) disturbance of impulse control, and (4) disturbance of social interaction. These scores a summed to a total score.

SECONDARY OUTCOMES:
total score for peer related aggression in the Questionnaire for Aggressive Behavior of Children (FAVK) teacher rating, patient self-report | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The Questionnaire for Aggressive Behavior of Children (FAVK) is a newly developed parent rating scale which assesses several factors of peer related aggression: (1) disturbance of social cognitive information processing, (2) disturbance of social problem solving and social skills, (3) disturbance of impulse control, and (4) disturbance of social interaction. These scores a summed to a total score. Self-report is assessed in children aged 9 or older.
ODD-Score of the Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV), parent, teacher and patient self-report | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV) assesses all symptom criteria for ODD and some of the symptom criteria of Conduct Disorders according to ICD-10 and DSM-IV. Self-report is assessed in children aged 11 or older.
ODD-Score of the Diagnostic Checklist for Oppositional Defiant and Conduct Disorder (DCL-SSV) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment)
  The Diagnostic Checklist for Oppositional Defiant and Conduct Disorder (DCL-SSV) is rated by a (blinded) clinician and assesses all symptom criteria for ODD and some of the symptom criteria of Conduct Disorders according to ICD-10 and DSM-IV based on parent information in a semi-structured interview.
Externalizing Problems Score of the Child Behavior Checklist (CBCL), the Teacher Report Form (TRF), and the Youth Self-Report (YSR) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The CBCL, TRF and YSR are well evaluated rating scales for the assessment of a broad spectrum of child behavioral and emotional problems as perceived by parents and teachers respectively. Self-report is assessed in children aged 11 or older.
Internalizing Problems Score of the Child Behavior Checklist (CBCL) and the Teacher Report Form (TRF) , and the Youth Self-Report (YSR) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The CBCL, TRF, and YSR are well evaluated rating scales for the assessment of a broad spectrum of child behavioral and emotional problems as perceived by parents and teachers respectively. Self-report is assessed in children aged 11 or older.
ADHD Symptom Checklist (FBB-ADHS) ,report parent, teacher and patient self-report ADHD Symptom Checklist (FBB-ADHS) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  ADHD Symptom Checklist (FBB-ADHS) assesses all symptom criteria for ADHD according to ICD-10 and DSM-IV. Self-report is assessed in children aged 11 or older.
ICU (Inventory of Callous-Unemotional Traits) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The ICU is designed to assess CU traits using self- and parent -report. The ICU consists of three subscales: Callousness, Uncaring and Unemotional. Self-report is assessed in children aged 9 or older
KINDL rating scale for quality of life, parent and patient self-report | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment)
  The KINDL is a German parent and patient rating scale for the assessment of different aspects of QoL. Self-report is assessed in children aged 7 or older.
FABEL rating scale for family burden | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment)
  The Modified FABEL is a parent rating scale for the assessment of different aspects of Family burden
Harter rating scale for self-concept | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The Modified Harter scale is a self rating scale for the assessment of different aspects of self-concept. Self-report is assessed in children aged 9 or older
Modified WFIRS (Weiss Functional Impairment Rating Scale) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment)
  The modified WFIRS is a parent rating scale for the assessment of psychosocial functioning in children with ODD/CD. The original WFIRS has been developed to assess psychosocial functioning in children with ADHD. Several items have been adapted or deleted in this modified version.
Individual Problem Checklist (IPC) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment)
  The IPC assesses individual problems as defined together with the parents. It represents the individual problems which were aimed to reduce with the treatment.
ScouT-Social Problem Solving Test (ScouT-SPST) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment)
  The ScouT-Social Problem Solving Test (ScouT-SPST) is a test that assesses problem solving compentecies according to the social problem solving theory (Dodge) as well as behavioural tendencies in specific conflict situations.
Depression Anxiety and Stress Questionnaire (DASS) | change from pre- to post1-assessment (24 weeks after pre-assessment), from post1- to post2-assessment (16 weeks after post1-assessment), and to follow up (12 months after post2-assessment)
  The DASS assesses parental depression anxiety and stress

CONTACTS AND LOCATIONS:
Overall Officials: Anja Goertz-Dorten, PhD, Principal Investigator — Department of Child and Adolescent Psychiatry Univ. Cologne
Locations (1):
- Department of Child and Adolescent Psychiatry at the University Cologne, Cologne, Germany

REFERENCES:
- [Derived] Goertz-Dorten A, Dose C, Hofmann L, Katzmann J, Groth M, Detering K, Hellmann A, Stadler L, Braun B, Hellmich M, Doepfner M. Effects of Computer-Assisted Social Skills Training in Children With Disruptive Behavior Disorders: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2022 Nov;61(11):1329-1340. doi: 10.1016/j.jaac.2022.03.027. Epub 2022 Apr 6. PMID 35398192